CLINICAL TRIAL: NCT06867614
Title: Laparoscopic Versus Transvaginal Closure of the Vaginal Vault After Total Laparoscopic Hysterectomy - a Single Blinded Randomized Comparative Study
Brief Title: Laparoscopic Versus Transvaginal Closure of the Vaginal Vault After Total Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rowan Ashraf AbdelHady Sakr, Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: FMASU MS 34/2025
Record Dates: First submitted 2025-02-18; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Total Laparoscopic Hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal approach (Active Comparator): Closure of vaginal vault after delivery of the specimen by vaginal suturing
  Interventions: Procedure: Total laparoscopic hysterectomy
- Laparoscopic approach (Active Comparator): Closure of vaginal vault after delivery of the specimen by laparoscopic suturing
  Interventions: Procedure: Total laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Total laparoscopic hysterectomy — Removal of uterus and cervix by laparoscope

SUMMARY:
The goal of this clinical trial is to compare the laparoscopic and transvaginal closure techniques of the vaginal vault in patients who perform TLH, regarding the risk of vaginal vault hematoma and other complications as vaginal cuff infection and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult females consenting to do TLH all age groups with diagnoses of benign uterine conditions.
* Women who are non-obese (normal or overweight women with BMI range 18-29.9).
* Sexually active female.

Exclusion Criteria:

* Diagnosed cases of pelvic malignancy
* Diagnosed patients with Cervical intraepithelial neoplasia (CIN) or bacterial vaginosis (any infection should be treated)
* Obese patients.
* Patients currently undergoing treatment for any type of cancer
* Patients with coagulopathy, bleeding/clotting disorders
* Patients with any condition can impair wound healing: diabetes mellites, anemia, steroids
* Patients with a previous history of radiation and allergy to sutures
* Patients with clinically evident prolapse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Vaginal Vault hematoma | From 10 days postoperative to 30 days postoperative
  It will be assessed by examination and ultrasound

SECONDARY OUTCOMES:
Bleeding/spotting | From 10 days postoperative to 30 days postoperative
  I wil be assed by history and examination
Vaginal infection: | From 10 days postoperative to 30 days postoperative
  It will be assessed by history and examination
Vaginal prolapse | From 10 days postoperative to 30 days postoperative
  It will be assessed by history and examination
Vaginal cuff granulation | From 10 days postoperative to 30 days postoperative
  It will be assessed by examination and ultrasound
Sexual dysfunction | From 3 to 4 months post operative
  I will be assessed through Female Sexual Function Index (FSFI) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No